CLINICAL TRIAL: NCT05133323
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of Lu AG09222 for the Prevention of Migraine in Patients With Unsuccessful Prior Preventive Treatments
Brief Title: A Study With Lu AG09222 in Adults With Migraine Who Have Not Been Helped by Prior Preventive Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19678A
Record Dates: First submitted 2021-11-15; First posted 2021-11-24 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lu AG09222 High Dose (Experimental): Participants will receive a single high dose of Lu AG09222 by intravenous (IV) infusion.
  Interventions: Drug: Lu AG09222
- Lu AG09222 Low Dose (Experimental): Participants will receive a single low dose of Lu AG09222 by IV infusion.
  Interventions: Drug: Lu AG09222
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo matching to Lu AG09222 by IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AG09222 — Lu AG09222 will be administered per schedule specified in the arm.
  Arms: Lu AG09222 High Dose; Lu AG09222 Low Dose
Drug: Placebo — Placebo matching to Lu AG09222 will be administered per schedule specified in the arm.
  Arms: Placebo

SUMMARY:
Researchers are trying to learn whether a drug called Lu AG09222 can help prevent migraine headaches for people who have not been helped by other treatments that are used to prevent migraines.

People who join this trial have tried 2 to 4 other medications to prevent their migraines, but these medications have not helped them.

When the trial is over, researchers will use this information to find out if the number of migraine days decreased more for the participants who got either dose of Lu AG09222 than for the participants who got the placebo.

DETAILED DESCRIPTION:
Participants will be randomly allocated to one of 3 treatment groups: Lu AG09222 high dose, Lu AG09222 low dose, or placebo, in a ratio of 2:1:2.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant has a diagnosis of migraine as defined by International Classification of Headache Disorders Third Edition (ICHD-3) guidelines confirmed at the Screening Visit.
* The participant has a history of migraine onset at least 12 months prior to the Screening Visit.
* The participant has a migraine onset at ≤50 years of age.
* The participant has documented evidence of treatment failure in the past 10 years of at least 2 to 4 (maximum) different migraine preventive medications.

Key Exclusion Criteria:

* The participant has been previously dosed with an anti-pituitary adenylate cyclase-activating polypeptide (anti-PACAP) ligand-targeting antibody.
* The participant has confounding and clinically significant pain syndromes.
* The participant has a diagnosis of acute or active temporomandibular disorder.
* The participant has a history or diagnosis of confounding headaches.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (28):
- United States (3):
  - Excell Research - ClinEdge - PPDS, Oceanside, California
  - UNISON Clinical Trials (Shahram Jacobs md inc.), Sherman Oaks, California
  - Allied Biomedical Research Institute, Miami, Florida
- Czechia (9):
  - CCR Ostrava s.r.o., Ostrava, Moravskoslezský kraj
  - Mestska nemocnice Ostrava, p.o., Ostrava, Moravskoslezský kraj
  - CCR Czech, Pardubice, Pardubický kraj
  - CCR Prague s.r.o., Prague, Praha, Hlavní Mesto
  - Fakultni nemocnice u sv. Anny v Brne, Brno, South Moravian
  - NEUROHK, s.r.o., Choceň
  - FORBELI s.r.o., Prague
  - INEP Medical s.r.o., Prague
  - CLINTRIAL s.r.o., Prague
- Denmark (2):
  - Rigshospitalet Glostrup-Nordre Ringvej 57, Glostrup Municipality, Capital
  - Aarhus Universitetshospital, Aarhus N, Central Jutland
- Georgia (6):
  - Ltd Israel-Georgia Medical Research Clinic Helsicore, Tbilisi
  - Archangel St Michael Multiprofile Clinical Hospital Ltd, Tbilisi
  - Aversi Clinic LTD, Tbilisi
  - LTD MediClubGeorgia, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, Tbilisi
  - Ltd Multiprofile Clinic "Consilium Medulla", Tbilisi
- Poland (6):
  - Solumed SC, Poznan, Greater Poland Voivodeship
  - Pratia MCM, Krakow, Lesser Poland Voivodeship
  - Instytut Zdrowia Dr Boczarska-Jedynak, Oświęcim, Lesser Poland Voivodeship
  - ETG Singua - PPDS, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Silmedic Sp z o o, Katowice, Silesian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw
- Slovakia (2):
  - MUDr. Beata Dupejova, Neurologicka ambulancia, s.r.o., Banská Bystrica
  - KONZILIUM s.r.o, Dubnica nad Váhom

REFERENCES:
- [Derived] Ashina M, Phul R, Khodaie M, Lof E, Florea I. A Monoclonal Antibody to PACAP for Migraine Prevention. N Engl J Med. 2024 Sep 5;391(9):800-809. doi: 10.1056/NEJMoa2314577. PMID 39231342

RESULTS

PARTICIPANT FLOW:
Groups:
- Lu AG09222 High Dose: Participants received a single dose of Lu AG09222 by intravenous (IV) infusion.
- Lu AG09222 Low Dose: Participants received a single dose of Lu AG09222 by IV infusion.
- Placebo: Participants received a single dose of placebo matching to Lu AG09222 by IV infusion.
Period: Overall Study
Arm/Group | Lu AG09222 High Dose | Lu AG09222 Low Dose | Placebo
Started | 97 | 46 | 94
Received at Least 1 Dose of Study Drug | 97 | 46 | 94
Completed | 95 | 45 | 93
Not Completed | 2 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The all-participants-treated set (APTS) represents all randomized participants who received an infusion of investigational medicinal product
Groups:
- Total: Total of all reporting groups
Arm/Group | Lu AG09222 High Dose | Lu AG09222 Low Dose | Placebo | Total
Number analyzed (Participants) | 97 | 46 | 94 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (9.88) | 42.5 (9.35) | 42.5 (9.51) | 42.5 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 38 | 81 | 208
  Male | 8 | 8 | 13 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 97 | 46 | 94 | 237
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Monthly Migraine Days (MMDs)
Description: The Migraine Day definition was based on the International Headache Society (IHS) guidelines for controlled trials of preventive treatment of chronic migraine and episodic migraine in adults. A Migraine Day was defined as a day with a headache that:
  * lasts ≥4 hours and meets International Classification of Headache Disorders Third Edition (ICHD-3) guidelines criteria C and D for migraine without aura
  * or lasts ≥30 minutes and where the participant had an aura with the headache (migraine with aura),
  * or lasts ≥30 minutes and meets two of the three ICHD-3 criteria B (without the condition on 72 hours), C and D for migraine without aura (probable migraine),
  * or a day with a headache that is successfully treated with a triptan, ergotamine, or other migraine-specific acute medication
Time Frame: Baseline, Week 4
Population: The APTS represents all randomized participants who received an infusion of investigational medicinal product
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Lu AG09222 High Dose | Lu AG09222 Low Dose | Placebo
Number analyzed (Participants) | 97 | 46 | 94
days | -6.2 (0.66) | -6.0 (0.94) | -4.2 (0.67)
Statistical Analysis 1: Comparison: Lu AG09222 High Dose vs Placebo; Test type: Superiority; p = 0.0106, ANCOVA; Mean Difference (Final Values) = -2.0, 90% CI 1-sided [upper limit -0.6], Standard Error of Mean 0.89

2. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in MMDs
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: The APTS represents all randomized participants who received an infusion of investigational medicinal product
Measure: Number; unit: percentage of participants
Arm/Group | Lu AG09222 High Dose | Lu AG09222 Low Dose | Placebo
Number analyzed (Participants) | 97 | 46 | 94
percentage of participants | 32.2 | 36.1 | 26.8

3. Secondary Outcome: Change From Baseline in the Number of Monthly Headache Days (MHDs)
Description: A Headache Day was defined as a day with a headache that lasted ≥30 minutes or that meets the definition of a Migraine Day.
Time Frame: Baseline, Week 4
Population: The APTS represents all randomized participants who received an infusion of investigational medicinal product. Here, 'Number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Lu AG09222 High Dose | Lu AG09222 Low Dose | Placebo
Number analyzed (Participants) | 96 | 44 | 93
days | -5.8 (0.65) | -5.9 (0.93) | -4.1 (0.67)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: The APTS represents all randomized participants who received an infusion of investigational medicinal product
Arm/Group | Lu AG09222 High Dose | Lu AG09222 Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/46 | 0/94
Serious Adverse Events (participants affected / at risk) | 1/97 | 0/46 | 0/94
Other Adverse Events (participants affected / at risk) | 18/97 | 4/46 | 8/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lu AG09222 High Dose (N=97) | Lu AG09222 Low Dose (N=46) | Placebo (N=94)
Sympathetic Posterior Cervical Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lu AG09222 High Dose (N=97) | Lu AG09222 Low Dose (N=46) | Placebo (N=94)
Covid-19 (Infections and infestations) | 7 (7) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 7 (7) | 0 (0) | 4 (5)
Fatigue (General disorders) | 5 (5) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT05133323/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT05133323/SAP_001.pdf